CLINICAL TRIAL: NCT02440724
Title: The Usefulness of Self-expandable Metal Stents(SEMS) for Malignant Gastric Outlet Obstruction: a Prospective Study Using New Designed Stents
Acronym: SEMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Yong Ahn, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0820
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Malignant Gastric Outlet Obstruction
Keywords: winged stents; Self-expandable Metal Stents(SEMS); partial covered; uncovered; endoscopic insertion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- winged stent group (Experimental): participants who are assigned to winged-stent group will be treated with deployment of a winged stent(partially covered or uncovered SEMS).
  Interventions: Device: Winged stent (partially covered); Device: Winged stent (uncovered)

INTERVENTIONS:
Device: Winged stent (partially covered) — A winged stent is a newly designed self-expandable metal stents(SEMS). Partially covered, or uncovered winged stent will be placed via the endoscopic intervention for malignant gastric outlet obstruction.
Device: Winged stent (uncovered) — A winged stent is a newly designed self-expandable metal stents(SEMS). Partially covered, or uncovered winged stent will be placed via the endoscopic intervention for malignant gastric outlet obstruction.

SUMMARY:
The purpose of this study is to evaluate usefulness of new designed winged stent(SEMS).

ELIGIBILITY:
Inclusion Criteria:

1. Gastric outlet obstruction symptom
2. Diagnosis of gastric outlet obstruction by radiologist or endoscopist
3. Gastric outlet obstruction by malignant disease
4. Aged over 19
5. Informed consent

Exclusion Criteria:

1. Gastric outlet obstruction by benign disease or infectious disease
2. Could not endoscopic intervention by poor general condition
3. Refusal of patient

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Complication rate(stent migration and tumor ingrowth) of new designed winged stent | up to 16 weeks from stent insertion
  It will be assessed by a composite measure consisting of physical exam, ECOG PS, GOOSS and gastrointestinal imaging.

SECONDARY OUTCOMES:
Evaluate the technical success rate of SEMS insertion | up to 16 weeks from stent insertion
  It will be assessed by a composite measure consisting of physical exam, ECOG PS, GOOSS and gastrointestinal imaging.
Evaluate the clinical success rate of SEMS insertion | up to 16 weeks from stent insertion
  It will be assessed by a composite measure consisting of physical exam, ECOG PS, GOOSS and gastrointestinal imaging.
Difference of insertion time between previous stent insertion and new designed stent | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Ji Yong Ahn, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea